CLINICAL TRIAL: NCT02751034
Title: A Randomized, Multi-center, Double Blind, Intra-Individual Controlled, Active-controlled Clinical Trial to Evaluate the Efficacy and Safety of Injection With Neuramis® Deep Lidocaine as Compared to Restylane® PERLANE-L in Correction of Nasolabial Fold
Brief Title: Efficacy and Safety Evaluation Study of Neuramis® Deep Lidocaine in Correction of Nasolabial Fold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT_PRT_NLF02
Record Dates: First submitted 2015-04-21; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Nasolabial Fold
Keywords: Wrinkle Severity Rating Scale; Global Aesthetic Improvement Scale; Hyaluronic acid filler; filler; Nasolabial Fold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuramis® Deep Lidocaine (Experimental): Neuramis® Deep Lidocaine Hyaluronic Acid Gel and Lidocaine Hydrochlorid, total dose 1ml, single injection
  Interventions: Device: Neuramis® Deep Lidocaine
- Restylane® PERLANE-L (Active Comparator): Restylane® PERLANE-L Hyaluronic Acid Gel and Lidocaine Hydrochlorid, total dose 1ml, single injection
  Interventions: Device: Restylane® PERLANE-L

INTERVENTIONS:
Device: Neuramis® Deep Lidocaine — HA filler
  Arms: Neuramis® Deep Lidocaine
Device: Restylane® PERLANE-L — HA filler
  Arms: Restylane® PERLANE-L

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the study medical device, Neuramis® Deep Lidocaine and the control medical device, Restylane® PERLANE-L in correction of nasolabial folds

DETAILED DESCRIPTION:
This study is a multi-center, double blind, intra-individual controlled, active-controlled clinical trial.

Efficacy and Safety are evaluated at the appointed time at subject visit clinical site after Injecting medical device.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged between 30 and 70 years, inclusive
2. Subjects who want improvement of bilateral nasolabial folds that are rated as 3 or 4 points on Wrinkle Severity Rating Scale
3. Subjects with visually symmetrical bilateral nasolabial folds
4. Subjects who consent to abstain from wrinkle improvement treatment in the lower face (below the lower orbital rim) during this trial
5. Subjects who are capable of understanding and following instructions, and participating in the entire course of the trial
6. Subjects who voluntarily decide to participate in this trial and provide written consent in the Informed Consent Form

Exclusion Criteria:

1. Subjects who administered an anticoagulant (except for low-dose aspirin (100mg, up to 300mg/day) or equivalent) within 2 weeks prior to screening
2. Subjects who had face-lift, soft tissue augmentation, medium or deeper peeling, or dermal photo-rejuvenation on the lower face (lower orbital rim) for wrinkle improvement within 6 months prior to screening
3. Subjects who received treatment with calcium hydroxyapatite(CaHA) at the investigational medical device injection site within 1 year from screening
4. Subjects who have implanted a permanent expander prosthesis at the investigational medical device injection site, such as soft-form or silicon
5. Subjects with a scar or skin lesion at the investigational medical device injection site that may interfere with judgment of the treatment effect
6. Subjects with a history of anaphylaxis or severe complicated allergy or allergy to lidocaine or hyaluronic acid products
7. Subjects with a history of a hypertrophic scar or keloid
8. Subjects with a skin disease or wound infection at the investigational medical device injection site
9. Subjects who participated in another clinical trial within 30 days prior to screening
10. Pregnant or breastfeeding women or women of childbearing potential who are not using medically acceptable contraception or not consenting to practice birth control from screening to the end of trial
11. Subjects who are otherwise determined by the investigator as ineligible for this study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change on the Wrinkle Severity Rating Scale as evaluated by photograph raters using photographs | from baseline to 24 weeks

SECONDARY OUTCOMES:
Change on Wrinkle Severity Rating Scale as evaluated by an investigator | from baseline to 8, 16, 24 weeks
Proportion of subjects with a ≥ 1 point change on Wrinkle Severity Rating Scale as evaluated by an investigator | from baseline to 8, 16, 24 weeks
Change on Wrinkle Severity Rating Scale as evaluated by photograph raters using photographs | from baseline to 8, 16 weeks
Proportion of subjects with a ≥ 1 point change on Wrinkle Severity Rating Scale as evaluated by photograph raters | from baseline to 8, 16, 24 weeks
Proportion of subjects with a ≥ 1 point on Global Aesthetic Improvement Scale as evaluated by an investigator | 8, 16, 24 weeks after the injection
Proportion of subjects with a ≥ 1 point on Global Aesthetic Improvement Scale as evaluated by a subject | 8, 16, 24 weeks after the injection
Visual Analogue Scale as evaluated by a subject | at 15, 30, 45, 60 minutes after the injection
Vital signs, physical examination, laboratory tests and adverse events | from baseline to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hoon Kang, Principal Investigator — Catholic University St. Paul Hospital; BeomJoon Kim, Principal Investigator — Chung-Ang Univ. Medical Center
Locations (2):
- South Korea (2):
  - Catholic University St. Paul Hospital, Seoul, Dongdaemun-gu
  - Chung-Ang Univ. Medical Center, Seoul, Dongjak-gu

IPD SHARING:
Plan to Share IPD: No